CLINICAL TRIAL: NCT04949516
Title: Aspirin-free Therapy After Successful Percutaneous Coronary Intervention for Acute Coronary Syndrome: the MACT (Mono Antiplatelet and Colchicine Therapy) Pilot Study
Brief Title: Mono Antiplatelet and Colchicine Therapy
Acronym: MACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Seung-Yul Lee, Associate Professor, Wonkwang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WKUH 2021-06-004
Record Dates: First submitted 2021-06-17; First posted 2021-07-02 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Acute Coronary Syndrome; Drug-Eluting Stents
Keywords: Platelet Aggregation Inhibitors; Colchicine
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mono Antiplatelet and Colchicine Therapy (Experimental): Aspirin-free, single P2Y12 inhibitor (prasugrel or ticagrelor) and colchicine treatment
  Interventions: Drug: Aspirin; Drug: Colchicine

INTERVENTIONS:
Drug: Aspirin — Aspirin is discontinued the day after drug-eluting stent implantation
  Other Names: Aspirin stop
Drug: Colchicine — Colchicine is started the day after drug-eluting stent implantation
  Other Names: Colchicine start

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of aspirin-free, P2Y12 inhibitor single antiplatelet and colchicine treatment in patients with acute coronary syndrome treated with drug-eluting stents.

DETAILED DESCRIPTION:
After successful drug-eluting stent implantation for acute coronary syndrome, screening for study subject enrollment is performed. For those who submitted written informed consent, aspirin is stopped the day after the intervention, and colchicine 0.6mg once daily is started. The P2Y12 inhibitor, prasugrel or ticagrelor, for single antiplatelet therapy remains. For the duration of hospital stay, platelet reactivity using VerifyNow test and C-reactive protein are measured. Aspirin may be restarted at the discretion of the investigator based on results of the platelet function test. C-reactive protein is remeasured 30 days after the intervention. Clinical follow-up is performed 30 days and 90 days after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Successful PCI with drug-eluting stent for NSTE-ACS or STEMI
* Provision of written informed consent

Exclusion Criteria:

* Cardiac arrest or cardiogenic shock
* Age <19 or >90 years old
* Severe liver impairment
* Severe renal impairment (eGFR <30 mL/min/1.73 m2)
* Atrial fibrillation requiring anticoagulation therapy
* Intolerance of prasugrel, ticagrelor, or colchicine
* History of intracranial hemorrhage
* Active bleeding

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes - Definite, probable, and possible stent thrombosis (Academic Research Consortium) | Assessed at hospital stay and 30/90 days after stent implantation
  Definite, probable, and possible stent thrombosis (Academic Research Consortium)

SECONDARY OUTCOMES:
Clinical outcomes - Target vessel failure | Assessed at hospital stay and 30/90 days after stent implantation
  Composite time-to-first event rate of cardiac death, target vessel-myocardial infarction (TV-MI), or ischemia driven-target vessel revascularization (ID-TVR)
Clinical outcomes - Target lesion failure | Assessed at hospital stay and 30/90 days after stent implantation
  Composite time-to-first event rate of cardiac death, TV-MI, or ischemia driven-target lesion revascularization (ID-TLR)
Clinical outcomes - All-cause mortality | Assessed at hospital stay and 30/90 days after stent implantation
  All-cause mortality
Clinical outcomes - Cardiac and non-cardiac mortality | Assessed at hospital stay and 30/90 days after stent implantation
  Cardiac and non-cardiac mortality
Clinical outcomes - All myocardial infarction | Assessed at hospital stay and 30/90 days after stent implantation
  All myocardial infarction
Clinical outcomes - TV-MI and non-TV-MI | Assessed at hospital stay and 30/90 days after stent implantation
  TV-MI and non-TV-MI
Clinical outcomes - All revascularization | Assessed at hospital stay and 30/90 days after stent implantation
  All revascularization
Clinical outcomes - ID-TVR, ID-TLR and ID-non-TLR TVR | Assessed at hospital stay and 30/90 days after stent implantation
  ID-TVR, ID-TLR and ID-non-TLR TVR
Clinical outcomes - Type 1, type 2, type 3, type 4, and type 5 bleeding (Bleeding Academic Research Consortium) | Assessed at hospital stay and 30/90 days after stent implantation
  Type 1, type 2, type 3, type 4, and type 5 bleeding (Bleeding Academic Research Consortium)
Laboratory outcomes - P2Y12 reaction unit | Assessed at hospital stay
  P2Y12 reaction unit using VerifyNow P2Y12 rapid analyzer
Laboratory outcomes - Percent platelet inhibition | Assessed at hospital stay
  Percent platelet inhibition using VerifyNow P2Y12 rapid analyzer
Laboratory outcomes - C-reactive protein | Assessed at hospital stay and 30 days after stent implantation
  C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yul Lee, MD, Principal Investigator — Wonkwang University Hospital
Locations (1):
- Wonkwang University Hospital, Iksan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SY, Cho JY, Gorog DA, Angiolillo DJ, Yun KH, Ahn JH, Koh JS, Park Y, Hwang SJ, Hwang JY, Kim JW, Jang Y, Jeong YH. Inflammation and platelet reactivity during adjunctive colchicine versus aspirin in patients with acute coronary syndrome treated with potent P2Y12 inhibitor. Front Med (Lausanne). 2024 Apr 19;11:1349577. doi: 10.3389/fmed.2024.1349577. eCollection 2024. PMID 38841588
- [Derived] Lee SY, Jeong YH, Yun KH, Cho JY, Gorog DA, Angiolillo DJ, Kim JW, Jang Y. P2Y12 Inhibitor Monotherapy Combined With Colchicine Following PCI in ACS Patients: The MACT Pilot Study. JACC Cardiovasc Interv. 2023 Aug 14;16(15):1845-1855. doi: 10.1016/j.jcin.2023.05.035. PMID 37587591